CLINICAL TRIAL: NCT06620445
Title: Efficacy of Psychological Intervention for Children With Cancer: A Randomized Controlled Trail
Brief Title: Efficacy of Psychological Intervention for Children With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Dr. Muhammad Wasim Khan, Dr. Muhammad Wasim Khan, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F.1-1/2015/ERBSZABMU/1311
Record Dates: First submitted 2024-09-10; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Clinical Depression; Clinical Anxiety; Quality of Life
Keywords: Psychological Intervention; Pediatric Cancer
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms

STUDY DESIGN:
Intervention Model Description: This single-blinded, two-arm randomized controlled trial will involve 80 children aged 8-16 with malignancies receiving chemotherapy.
  Participants will be randomly assigned to either the experimental group, which will receive five weekly sessions of cognitive-behavioral intervention, or the control group, which will receive usual care. Each intervention session will last 30-35 minutes.
  Outcomes will be measured at baseline and one-month post-intervention using the Revised Child Anxiety and Depression Scale and Pediatric Quality of Life Inventory Generic Core Score 4.0.
Who Masked: Participant
Masking Description: Participants (Children/Guaddians or Parents) are unaware of which group they are assigned (CBT group or usual care group). Researcher are aware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): The Intervention or CBT group included 40 children aged 8-16 years with malignancies recieving chemotherapy. They will recieve weekly five sessions of CBT (30-35 minutes per session)
  Interventions: Behavioral: Interventiion or CBT Group
- Control or Usual Care Group (No Intervention): The Control or No Intervention Group also known as Comparision Group or Usual Group will recieve the standard care or usual care for their condition. It will serve as a baseline for the CBT or Intervention Group.

INTERVENTIONS:
Behavioral: Interventiion or CBT Group — This RCT aims to evaluate the effect of Cognitive Behavioral Therapy (CBT) compared to usual care (UC) in pediatric oncology patients. We hypothesize that those receiving CBT will report lower depression and anxiety and improved QoL six months post-enrollment.
  Other Names: Cognitive or Pschological Intervention
  Arms: Interventional Group

SUMMARY:
The study will be conductued at the Pediatric Oncology Department of the Children's Hospital, PIMS Islamabad, over the peroid of six months. This single-blinded, two-arm RCT study will involve 80 children aged 8 to 16 years with maligancies recieving chemotherapy. Participants will be randomly allocated to either interventional or CBT group which will recieve weekly five sessions of Cognitive Behaviour Therapy (CBT) or the control group, which will recieve the usual care. CBT session will be contducted by Clinical Psychologist will last 30-35 minutes. Outcomes will be measured at Baseine and one month post intervention using Revised Child Anxiety and Depression Scale (RCADS) and Pediatric Quality of Life Generic Core Score 4.0.

DETAILED DESCRIPTION:
Background:

Children with cancer and their families experience various psychosocial challenges during and after treatment, including physical and cognitive changes due to medical treatment, alterations in social and familial roles, and the potential threat of death.

While most children and families cope and adjust well to the diagnosis and treatment of cancer, a subset of children is at increased risk for anxiety, depression, educational, and relationship difficulties. Caregivers and siblings of pediatric patients are also at risk for heightened distress and post-traumatic stress. Psychosocial care and interventions can play an important role in supporting the well-being of the entire family, beginning at diagnosis.

The psychological impact of cancer on Pakistani children is diverse and far-reaching, ranging from concerns about their future to worries about appearing different from their peers. Given the high prevalence of psychological difficulties among pediatric cancer patients in Pakistan, it is essential to determine the effectiveness of interventions offered to support their mental health and well-being. Studies on cancer patients related to their psychiatric problems are already rare in Pakistan.

Objective:

The main objective of this study is to compare the effect of psychological intervention, such as cognitive-behavioral therapy (CBT), to the routine care given among pediatric oncology patients. The findings of this study will provide evidence to support the integration of psychological intervention strategies into pediatric oncology practice, thus adding new knowledge to the literature and helping improve the care of children with malignancies receiving chemotherapy.

Study Design:

The study will be conducted at the Pediatric Oncology Unit, PIMS, Islamabad. This study will be a two-armed longitudinal, randomized control trial expected to run for six months. Children with malignancy receiving chemotherapy will be recruited and randomly assigned to experimental or control groups.

Intervention:

The experimental group will receive five sessions of cognitive-behavioral intervention, where maladaptive thoughts and behavior will be identified, behavioral activation will be encouraged, and deep breathing exercises will be practiced. The control group will receive the usual care.

Recruitment and Sample:

The recruitment process will involve the random selection of children diagnosed with malignancies and undergoing treatment at the Pediatric Oncology Unit, the Children's Hospital PIMS Islamabad, Pakistan.

Outcome Measures:

The outcomes will be measured at baseline, post-intervention, and one month after the intervention using the Revised Child Anxiety and Depression Scale and Pediatric Quality of Life Inventory Generic Core Score 4.0.

Data Analysis:

Data analysis will be conducted using SPSS version 23.

Ethical Considerations:

Permission to conduct the study will be acquired from the Ethical Review Board (ERB) of PIMS Islamabad.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

1. Children aged 16-18 years
2. Diagnosed with malignancy
3. Recieving chemotherapy at the Pediatric Oncology Department of PIMS Islamabad
4. Able to understand and participate in CBT sessions
5. Parent/Caregiver consent and child assent

Exlusion Criteria:

1. Children with severe cognitive impairment or intellectual disability
2. Children with a comorbid medical conditions
3. Children whose parents or caregivers are unable to provide consent

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS) | Baseline (before the intervention) and one month post intervention (after the five weekly sessions of CBT)
  The RCADS is a standardized, self reported scale measuring anxiety and depression symptoms among children aged 8-18 years.

SECONDARY OUTCOMES:
Pediatric QoL | Baseline and one month post intervention
  It evaluates physical, emotional, social and school funtioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammad Wasim Khan, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
Demographic, Clinical and Treatment related Information of the Participants

DOCUMENTS (3):
  • Study Protocol (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT06620445/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT06620445/SAP_001.pdf
  • Informed Consent Form (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT06620445/ICF_002.pdf